CLINICAL TRIAL: NCT06787638
Title: Diaphragmatic Dynamics in Laparoscopic Cholecystectomy: Comparing Neuromuscular Blocker Reversal Strategies-A Randomized Trial
Brief Title: Effects of Neostigmine-dose on Diaphragmatic Dynamics
Acronym: DTF/DE/AChE
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Sara Abd El Dayem Mohamed Abed, Resident of anesthesia, surgical intensive care & pain management, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 944/7/24
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Diaphragm Ultrasound
Keywords: Diaphragmatic Thickening Fraction; Diaphragmatic Excursion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- full dose of Neostigmine (Active Comparator)
  Interventions: Drug: full dose of Neostigmine
- half dose of Neostigmine (Active Comparator)
  Interventions: Drug: half dose of Neostigmine

INTERVENTIONS:
Drug: full dose of Neostigmine — • Group A: received 10ml (a full dose of Neostigmine (0.08 mg/kg) plus Atropine (20 mic/kg+7ml normal saline)
  Measured using ultrasound Time frame: preoperatively and at zero, 10 minutes and 30 minutes postoperatively.
  Arms: full dose of Neostigmine
Drug: half dose of Neostigmine — • Group B: received 10ml (a half dose of Neostigmine (0.04 mg/kg) plus Atropine (20 mic/kg+8ml normal saline).
  Measured using ultrasound Time frame: preoperatively and at zero, 10 minutes and 30 minutes postoperatively.
  Arms: half dose of Neostigmine

SUMMARY:
The goal of this Randomized Clinical Trial is to compare the postoperative diaphragmatic excursion between patients receiving half-dose neostigmine (0.04 mg/kg) and those receiving full-dose neostigmine (0.08 mg/kg) for neuromuscular blockade reversal.

The main questions it aims to answer are:

* Does half-dose neostigmine result in similar postoperative diaphragmatic excursion compared to full-dose neostigmine?
* Does half-dose neostigmine result in similar diaphragmatic thickening fraction compared to full-dose neostigmine? Researchers will compare patients receiving half-dose neostigmine to those receiving full-dose neostigmine to see if there are differences in postoperative diaphragmatic function, respiratory complications, and recovery.

Participants will:

* Undergo elective laparoscopic cholecystectomy.
* Receive either half-dose or full-dose neostigmine for neuromuscular blockade reversal.

DETAILED DESCRIPTION:
Fifty patients from both genders scheduled for elective laparoscopic cholecystectomy were enrolled in this study to compare diaphragmatic assessment parameters.

Enrolled participants were randomly assigned to group A (patient receiving full dose of Neostigmine (0.08 mg/kg) plus Atropine (20 mic/kg)) or group B (patient receiving half dose of Neostigmine (0.04 mg/kg) plus Atropine (20 mic/kg)).

This is a prospective study that will be conducted at Aswan University Hospital.

Eligible participants will be adult patients (age ≥ 18 years) scheduled for elective laparoscopic cholecystectomy, with American Society of Anesthesiologists (ASA) physical status I or II, and a body mass index (BMI) < 35 kg/m². Patients with pre-existing diaphragmatic or respiratory disorders, ASA physical status III or IV, BMI > 35 kg/m², chronic opioid use or abuse, pregnancy, or breastfeeding will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Adults scheduled for elective laparoscopic cholecystectomy.
* Age: < or = 18 years.
* Both genders.
* American Society Of Anesthiologists (ASA) I/II patients.
* BMI <35

Exclusion Criteria:

* Pre-existing diaphragmatic or respiratory disorders.
* ASA III/IV
* BMI >35
* Chronic opioid use or abuse
* Pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-25 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic Dynamics | preoperatively and at zero, 10 minutes and 30 minutes postoperatively
  To compare the postoperative diaphragmatic excursion between patients receiving half-dose neostigmine (0.04 mg/kg) and those receiving full-dose neostigmine (0.08 mg/kg) for neuromuscular blockade reversal.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman M El-demirdash, Study Chair — Anesthesia, surgical intensive care and pain management - Aswan University Hospital; Hani M Raslan, Study Director — Anesthesia, surgical intensive care and pain management - Aswan University Hospital; Zaher Z Zaher, Study Director — Anesthesia, surgical intensive care and pain management - Aswan University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayoub J, Cohendy R, Prioux J, Ahmaidi S, Bourgeois JM, Dauzat M, Ramonatxo M, Prefaut C. Diaphragm movement before and after cholecystectomy: a sonographic study. Anesth Analg. 2001 Mar;92(3):755-61. doi: 10.1097/00000539-200103000-00038. PMID 11226114
- [Background] Alam MJ, Roy S, Iktidar MA, Padma FK, Nipun KI, Chowdhury S, Nath RK, Rashid HO. Diaphragm ultrasound as a better predictor of successful extubation from mechanical ventilation than rapid shallow breathing index. Acute Crit Care. 2022 Feb;37(1):94-100. doi: 10.4266/acc.2021.01354. Epub 2022 Jan 11. PMID 35081706
- [Background] Adeyinka A, Layer DA. Neuromuscular Blocking Agents. 2024 Jun 8. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK537168/ PMID 30725853